CLINICAL TRIAL: NCT02123173
Title: Hemodynamic Changes and Fluid Responsiveness During One Lung Ventilation: Comparison in Non-intubated and Intubated Vedio-assisted Thoracoscopic Operations
Brief Title: Hemodynamic Changes During One Lung Ventilation in Non-intubated Vedio-assisted Thoracoscopic Operations
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201401037RINB
Record Dates: First submitted 2014-04-21; First posted 2014-04-25 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Lung Neoplasms
Keywords: one lung ventilation,; cardiac output; fluid responsiveness
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- non-intubated: VATS, non-intubated
- intubated: VATS, intubated

SUMMARY:
Non-intubated thoracoscopic surgery has been proved as an adequate alternative for management of many lung conditions such as pneumothorax , lung volume reduction, pulmonary metastasectomy, removal of lung nodules, segmentectomy and lobectomy. However, the hemodynamic changes during one lung ventilation have not been fully investigated. The goals of this study are to compare the changes of hemodynamics (including blood pressure, heart rate, cardiac output, pulse pressure variation, fluid responsiveness) during one lung ventilation between conventional intubated and non-intubated vedio-assisted thoracoscopic (VATS) operations.

DETAILED DESCRIPTION:
Non-intubated vedio-assisted thoracoscopic (VATS) is proved safely performed as well as traditional intubated VATS. However, the differences of hemodynamic changes and fluid responsiveness during one lung ventilation(OLV) between these two groups were rarely reported. For complete lung collapse, spontaneous negative pressure respiration must be well maintained on non-intubated VATS. In comparison, positive pressure ventilation on dependent lung was applied during OLV in intubated VATS. This study planned to compared the changes of hemodynamics (including blood pressure, heart rate, cardiac output) during OLV between groups. As functional hemodynamic monitoring (FloTrac system) was mostly utilized with positive pressure ventilation, the applicability of FloTrac in non- intubated VATS was also testified. In this study, we also measure the fluid responsiveness by FloTrac system with rapid infusion (within 10 minutes) of 10 mL/kg crystalloid fluid. We planned to compare the changes on cardiac output and the fluid responsiveness during OLV between these two groups.

ELIGIBILITY:
Inclusion criteria:

1. age over 20 y/o, less than 70 y/o
2. scheduled to receive VATS operations with OLV

Exclusion:

1. previous thoracic surgery
2. cardiac disease ( including arrhythmias, congestive heart failure, coronary cardiac disease, etc.)
3. pulmonary disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled to receive video-assisted thoracoscopic (VATS) operations with one lung ventilation(OLV)
  Inclusion criteria:
  1. age over 20 y/o, less than 70 y/o
  2. scheduled to receive VATS operations with OLV
  Exclusion:
  1. previous thoracic surgery
  2. cardiac disease ( including arrhythmias, congestive heart failure, coronary cardiac disease, etc.)
  3. pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
cardiac output after one lung ventilation | 10-15 minutes
  record the stroke volume and cardiac output during two lung ventilation till 15 minutes after one lung ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Jung Cheng, Principal Investigator — department of anesthesiology, national taiwan university hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan